CLINICAL TRIAL: NCT06531824
Title: A Multicenter, International, Randomized, Double-blind, Placebo-controlled Clinical Trial of the Aldosterone Synthase Inhibitor BI 690517 in Combination With Empagliflozin in Patients With Chronic Kidney Disease
Brief Title: EASi-KIDNEY™ (The Studies of Heart & Kidney Protection With BI 690517 in Combination With Empagliflozin)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1378-0006; 2024-511025-63-00 (Registry Identifier: CTIS); U1111-1306-5049 (Registry Identifier: WHO register (ICTRP))
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Kidney Disease, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Part 1: Run-in period, non randomized, single arm Part 2: Randomized (BI 690517 or placebo), double-blind, placebo-controlled follow-up period
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Run-in period (all participants) (Other): Eligible participants will enter a Run-in period during which they will receive placebo matching BI 690517 + empagliflozin.
  Interventions: Drug: Placebo matching BI 690517; Drug: Empagliflozin
- Part 2: Randomized treatment, follow-up period, treatment group (Experimental)
  Interventions: Drug: BI 690517; Drug: Empagliflozin
- Part 2: Follow-up period, placebo group (Placebo Comparator)
  Interventions: Drug: Placebo matching BI 690517; Drug: Empagliflozin

INTERVENTIONS:
Drug: BI 690517 — BI 690517
  Other Names: Vicadrostat
  Arms: Part 2: Randomized treatment, follow-up period, treatment group
Drug: Placebo matching BI 690517 — Placebo matching BI 690517
  Arms: Part 1: Run-in period (all participants); Part 2: Follow-up period, placebo group
Drug: Empagliflozin — Empagliflozin

SUMMARY:
This study is open to adults with chronic kidney disease at risk of progression. People with and without type 2 diabetes can take part in this study. The study is open to people who take other medicines called angiotensin converting enzyme inhibitors (ACEi) or angiotensin receptor blockers (ARB). People who already take empagliflozin or any other sodium-glucose cotransporter-2 inhibitor (SGLT2i) can also join. The study is also open to people who currently do not take any of these treatments. The purpose of this study is to find out whether a medicine called BI 690517 helps people with chronic kidney disease when taken in combination with a study medicine called empagliflozin. Worsening of kidney function increases the risk for kidney failure, cardiovascular disease, and heart disease.

This study has 2 parts. In the first part, participants get empagliflozin or placebo matching BI 690517 for at least 6 weeks. Participants continue taking ACEi or ARB throughout the study if such treatments are indicated. In the second part, participants are divided into 2 groups by chance. One group takes BI 690517 tablets and the other group takes placebo tablets. Placebo tablets look like BI 690517 tablets but do not contain any medicine. Participants take 1 tablet once a day in addition to empagliflozin for the duration of the study.

The doctors document when participants experience worsening of their kidney disease, go to hospital due to heart failure, or die of cardiovascular problems during the study. The time to these events is compared between the 2 treatment groups to see whether the treatment works. The study continues until the required number of events have occurred which is about 3 to 4 years. During this time, participants visit the study site about 4 times within the first 6 months. Then they visit the study site every 6 months. At the visits, doctors regularly check participants' health, take blood and urine samples, measure blood pressure and weight, check kidney function, and take note of any unwanted effects.

ELIGIBILITY:
Key Inclusion Criteria:

* Evidence of chronic kidney disease (CKD) at risk of kidney disease progression is defined on the basis of local laboratory results recorded at least 3 months before and at the time of the Screening visit, and requires:

  1. Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) eGFR ≥20 <45 mL/min/1.73m²; or
  2. CKD-EPI eGFR ≥45 <90 mL/min/1.73m² with urine albumin-to-creatinine ratio (uACR) ≥200 mg/g (or protein-to-creatinine ratio ≥300 mg/g).
* Neither requires an Aldosterone Synthase inhibitor (ASi) or Mineralocorticoid Receptor Antagonist (MRA), nor that such treatment is definitely inappropriate.

Key Exclusion Criteria:

* Blood potassium of >5.2 mmol/L at screening visit
* Blood Alanine Transaminase (ALT) or Aspartate Transaminase (AST) >3x Upper Limit of Normal (ULN) at Screening visit
* Known liver cirrhosis
* On dialysis, functioning kidney transplant, or scheduled living donor transplant
* Treated with new immunosuppression therapy for new (or relapse/flare of pre-existing) kidney disease within the last 60 days
* Receiving more than one Renin-Angiotensin System (RAS) inhibitor (i.e. on dual therapy with two of an Angiotensin-Converting Enzyme inhibitor (ACEi), Angiotensin Receptor Blocker (ARB) or direct renin inhibitor)
* Currently treated with an Mineralocorticoid Receptor Antagonist (MRA) (e.g. spironolactone, eplerenone, finerenone)
* Currently treated with systemic mineralocorticoid replacement therapy (e.g. fludrocortisone) Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11000 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2028-08-30 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
Time to first occurrence of the primary composite outcome of: (i) Kidney disease progression*; or (ii) Hospitalization for heart failure; or (iii) Cardiovascular death. | up to 4 years
  Kidney disease progression is defined as kidney failure or a sustained decline of ≥40% in estimated Glomerular Filtration Rate (eGFR) from randomization

SECONDARY OUTCOMES:
Key secondary outcome: Annual rate of change in eGFR from 3 month visit until last scheduled visit (i.e. chronic eGFR slope) | up to 4 years
Time to first event of kidney failure, hospitalization for heart failure or cardiovascular death | up to 4 years
Time to kidney disease progression | up to 4 years
Occurrences of hospitalizations for heart failure (first and any subsequent, combined) or cardiovascular death | up to 4 years
Occurrences of hospitalizations from any cause (first and any subsequent, combined) | up to 4 years
Time to first event of kidney disease progression or cardiovascular death | up to 4 years
Time to death from any cause | up to 4 years

CONTACTS AND LOCATIONS:
Locations (346):
- United States (24):
  - Apogee Clinical Research, Huntsville, Alabama
  - Southwest Kidney Institute, Surprise, Arizona
  - Florida Kidney Physicians LLC, Jacksonville Beach, Florida
  - Total Research Group, LLC, Miami, Florida
  - East Coast Institute For Research LLC, Macon, Georgia
  - Kootenai Research Services, Coeur d'Alene, Idaho
  - Kansas Nephrology Research Institute, LLC, Wichita, Kansas
  - Lake Michigan Nephrology, Saint Joseph, Michigan
  - St. Clair Nephrology Research, LLC, Shelby, Michigan
  - Great Plains Nephrology, North Platte, Nebraska
  - Sierra Nevada Specialty Care, Reno, Nevada
  - Seacoast Kidney and Hypertension Specialists, Portsmouth, New Hampshire
  - Metrolina Nephrology Associates, PA, Charlotte, North Carolina
  - Brookview Hills Research Associates LLC, Winston-Salem, North Carolina
  - Northeast Endocrine Metabolic Associates, Philadelphia, Pennsylvania
  - Clinical Renal Associates, Upland, Pennsylvania
  - Nephrology Associates, Inc, East Providence, Rhode Island
  - Dallas Nephrology Associates Medical Clinic, DeSoto, Texas
  - P&I Clinical Research, LLC, Lufkin, Texas
  - Texas Institute for Kidney and Endocrine Disorders, Lufkin, Texas
  - Renal Specialists of Houston, PA, Pasadena, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Tidewater Physicians Multispecialty Group, Newport News, Virginia
  - Providence Medical Research Center, Spokane, Washington
- Argentina (15):
  - Fundacion INTECNUS, Bariloche
  - Centro de Salud Renal Junín SRL, Buenos Aires
  - Dres. Iribarren & Asoc. Consultario, Buenos Aires
  - Glenny Corp - Centro Médico Saavedra, Buenos Aires
  - Sanatario Pasteur, Catamarca
  - CIMEL Chahin - Chahin S.A., Lanús Este
  - Mains Bleues, Rafaela
  - Hospital Privado de Rosario, Rosario
  - Sanatorio Parque S.A., Rosario
  - Instituto de Nefrourología y Nutrición de Salta, Salta
  - Clínica El Castaño, San Juan
  - Centro de Investigaciones Médicas Tucumán, San Miguel de Tucumán
  - Centro Integral de Medicina Respiratória - CIMER, San Miguel de Tucumán
  - Instituto de Investigaciones Clinicas de Rosario, Santa Fe
  - CEREHA S.A.- Centro de Estudios Renales e Hipertensión Arterial, Villa Domínico
- Australia (3):
  - Renal Research, Gosford, Gosford, New South Wales
  - Port Macquarie Base Hospital (PMBH), Port Macquarie, New South Wales
  - Sunshine Hospital, St Albans, Victoria
- Brazil (21):
  - Centro de Pesquisa Clínica do Coração, Aracaju
  - Centro de Pesquisa do Hospital Evangélico de Belo Horizonte, Belo Horizonte
  - Hospital Universitário São Francisco na Providência de Deus, Bragança Paulista
  - CEG - Centro de Endocrinologia Geloneze, Campinas
  - Instituto Cardiovascular de Linhares Ltda, Centro Linhares
  - Hospital Universitário Walter Cantídio - UFC, Fortaleza
  - Centro de Pesquisas em Diabetes e Doencas Metabolicas, Fortaleza
  - Clínica CENDI Endocrinologia e Diabetes, Goiânia
  - Hospital Ruy Azeredo, Goiânia
  - Fundação Pró-Rim Joinville, Joinville
  - Galileo Medical Research Ltda, Juiz de Fora
  - Centro de Pesquisas Clínicas Dr. Marco Mota, Maceió
  - Hospital Universitário Onofre Lopes, Natal
  - IMIP Pernambuco, Recife
  - AME Saúde, Recife
  - Hospital das Clínicas da Universidade Federal de Pernambuco, Recife
  - Fundação Bahiana de Infectologia, Salvador
  - CIPES - Centro Internacional de Pesquisa Clínica, São José dos Campos
  - Instituto de Assistência Médica ao Servidor Público Estadual de São Paulo, São Paulo
  - Fundação Oswaldo Ramos (Hospital do Rim), São Paulo
  - Clínica Cardiológica, Votuporanga
- Canada (24):
  - University of Alberta Hospital (University of Alberta), Edmonton, Alberta
  - Royal Inland Hospital, Kamloops, British Columbia
  - Kelowna General Hospital, Kelowna, British Columbia
  - Northern Health, Prince George, British Columbia
  - Fraser Health, Surrey, British Columbia
  - St. Paul's Hospital (Vancouver), Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - CIUSSS Nord de l'île de Montreal, Québec, Montréal
  - Centre for Clinical Research, Halifax, Nova Scotia
  - Centricity Research (Brampton), Brampton, Ontario
  - Centricity Research (Vaughan), Concord, Ontario
  - Queen's University, Kingston, Ontario
  - London Regional Cancer Program - London Health Sciences Ctr., London, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - CIUSSS de l'Est-de-l'Île-de-Montréal, Montreal, Quebec
  - McGill University Health Centre (MUHC), Montreal, Quebec
  - CIUSSS de l Estrie-CHUS, Sherbrooke, Quebec
  - Centre hospitalier de l'Université de Montréal (CHUM), Montreal
  - CHU de Quebec-Universite Laval Research Centre, Québec
  - Diex Recherche Québec, Québec
- China (24):
  - Ansteel Group General Hospital, Anshan
  - Beijing AnZhen Hospital, Capital Medical University, Beijing
  - Fuwai Hospital, CAMS&PUMC, Beijing
  - The Second Hospital of Chaoyang, Chaoyang
  - Guangzhou Red Cross Hospital, Guangzhou
  - The Third Affiliated Hospital of Southern Medical University, Guangzhou
  - Guangdong Provincial Hospital of Chinese Medicine, Guangzhou
  - Shulan(Hanghzhou) Hospital, Hanghzhou
  - Zhejiang Hospital, Hangzhou
  - The Second Affiliated Hospital of Heilongjiang University of Chinese Medicine, Harbin
  - The Second People's Hospital of Hefei, Hefei
  - International Mongolian Hospital of Inner Mongolia, Hohot
  - Henan Jiyuan People's Hospital, Jiyuan
  - Luoyang Central Hospital, Luoyang
  - Jiangxi Branch Hospital of Xiangya Hospital of Central South University, Nanchang
  - Qingdao Cardiovascular Hospital, Qingdao
  - Shanghai Tenth People's Hospital, Shanghai
  - Shenzhen Nanshan People's Hospital, Shenzhen
  - Taizhou Hospital of Zhejiang Province, Taizhou
  - The Fourth Central Hospital of Tianjin, Tianjin
  - Xiamen Cardiovascular Hospital Xiamen University, Xiamen
  - Xinxiang Central Hospital, Xinxiang
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang
  - Zhuzhou Central Hospital, Zhuzhou
- Denmark (7):
  - Aalborg Universitetsshospital, Aalborg
  - Rigshospitalet, København, Copenhagen
  - Herlev and Gentofte Hospital, Herlev
  - Steno Diabetes Center Copenhagen, Herlev
  - Kolding Hospital, Kolding
  - Odense University Hospital, Odense
  - Zealand University Hospita; Roskilde, Roskilde
- Germany (45):
  - Universitätsklinikum Aachen, AöR, Aachen
  - Nephrologische Gemeinschaftspraxis Bad Nenndorf, Bad Nenndorf
  - Herz- und Diabeteszentrum Nordrhein-Westfalen, Bad Oeynhausen, Bad Oeynhausen
  - Praxis für Nierenkrankheiten und Dialyse Helle Mitte, Berlin
  - Universitätsklinikum Bonn AöR, Bonn
  - Städtisches Klinikum Braunschweig gGmbH, Braunschweig
  - KfH Nierenzentrum Coburg, Coburg
  - Klinikum Dortmund gGmbH, Dortmund
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Dialysezentrum Elsenfeld, Elsenfeld
  - ClinPhenomics CVC GmbH, Frankfurt
  - Agaplesion Markus Krankenhaus, Frankfurt am Main
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Nierenzentrum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Gießen und Marburg GmbH, Giessen
  - Universitätsklinikum Halle (Saale) AöR, Halle
  - Universitätsklinikum Hamburg, Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Zentrum Für Nieren Hochdruck und Stoffwechselerkrankungen, Hanover
  - BAG für Nephrologie und Dialyse, Heilbronn
  - Ruhr-Universität Bochum, Herne
  - Universität des Saarlandes, Homburg
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Klinikum Konstanz, Konstanz
  - KfH-Nierenzentrum Kronach, Kronach
  - Dr. Vehling-Kaiser MVZ GmbH, Landshut
  - KfH Nierenzentrum Leipzig, Leipzig
  - Nephrologisches Zentrum Emsland, Lingen
  - Universitätsklinikum Magdeburg AöR, Magdeburg
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Klinikum der Universität München - Campus Innenstadt, München
  - Klinikum rechts der Isar der Technischen Universität München, München
  - Dialysezentrum Neckarsulm, Neckarsulm
  - Universitätsklinikum Ruppin-Brandenburg, Neuruppin
  - Universitätsmedizin Rostock, Rostock
  - Dialysezentrum Rotenburg, Rotenburg (Wümme)
  - MVZ Dialysezentrum Schweinfurt, Schweinfurt
  - Städtisches Klinikum Solingen gGmbH, Solingen
  - Robert-Bosch-Krankenhaus GmbH, Stuttgart
  - KfH-Nierenzentrum Traunstein, Traunstein
  - Nephrologisches Zentrum Villingen-Schwenningen, Villingen-Schwenningen
  - Nierenzentrum Wiesbaden, Wiesbaden
  - Helios Universitätsklinikum Wuppertal, Wuppertal
  - Universitätsklinikum Würzburg AÖR, Würzburg
- India (27):
  - Manipal Hospital, Bangalore
  - St John's Medical College, Bangalore
  - Apollo Hospital - Bangalore, Bangalore
  - All India Institute of Medical Sciences Bhubaneswar, Bhubaneswar
  - Post Graduate Institute of Medical Education and Research, Chandigarh
  - Apollo Hospital - Chennai, Chennai
  - Karnataka Medical college and research institute, Hubballi
  - Osmania Medical College & Hospital, Hyderabad
  - Apollo Hospitals Jubilee Hills, Hyderabad
  - Apollo DRDO Hospital, Hyderabad
  - Amrita Institute of Medical Sciences and Research Centre, Kochi
  - Nil Ratan Sircar Medical College & Hospital, Kolkata
  - IQRAA International hospital & research centre., Kozhikode
  - Dr Ram Manohar Lohia Institute of Medical Sciences, Lucknow
  - Apollo Speciality Hospital, Madurai, K.K. Nagar
  - Apollo BGS Hospital, Mysore
  - Muljibhai Patel Urological Hospital, Nadiād
  - Max Super Specialty Hospital, Saket, New Delhi
  - Epitome Kidney Urology Institute and Lions Hospital, New Delhi
  - All India Institute of Medical Sciences, New Delhi
  - Fortis Flt. Lt. Rajan Dhall Hospital, New Delhi
  - Indira Gandhi Institute of Medical Sciences, Patna
  - Jawaharlal Institute of Postgraduate Medical Education, Puducherry
  - All India Institute of Medical Sciences, Raipur
  - Yashoda Hospitals - Secunderabad, Secunderabad
  - Kimshealth, Trivandrum
  - Christian Medical College, Vellore, Vellore
- Italy (28):
  - Ospedale Civile Ss. Antonio e Biagio, Alessandria
  - Asti-Ospedale Cardinal Massaia, Asti
  - Azienda Universitaria Ospedaliera Consorziale Policlinico Bari, Bari
  - ASST Papa Giovanni XXIII, Bergamo
  - Policlinico S. Orsola-Malpighi, Bologna
  - Azienda Ospedaliera ARNAS G. Brotzu, Cagliari
  - Chieri-Ospedale Maggiore, Chieri
  - A.S.O.S. Croce e Carle, Cuneo
  - Firenze-Ospedale San Giovanni di Dio, Florence
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Azienda Ospedaliera San Martino, Genova
  - Ospedale di Imola S. Maria della Scaletta, Imola
  - Asst Santi Paolo E Carlo, Milan
  - Fondazione IRCCS San Gerardo dei Tintori, Monza
  - Ospedale Maggiore della Carità, Novara
  - Azienda Ospedaliera Unversitaria di Parma, Parma
  - Fondazione Salvatore Maugeri, Pavia
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - Prato-Ospedale Santo Stefano, Prato
  - Azienda Ospedaliera Sant'Andrea-Università di Roma La Sapienza, Roma
  - Ospedale Sant'Anna di San Fermo della Battaglia, San Fermo della Battaglia
  - IRCCS Ospedale "Casa Sollievo della Sofferenza", San Giovanni Rotondo (Foggia)
  - Azienda Sociosanitaria Ligure 2, Savona
  - IRCCS MultiMedica, Sesto San Giovanni
  - Todi-Nuovo Ospedale Media Valle del Tevere, Todi
  - Torino-Ospedale Oftalmico, Turin
  - Ospedale Castelli - Verbania, Verbania
  - Ospedale San Bortolo, Vicenza
- Japan (13):
  - University of Yamanashi Hospital, Chuo-Shi
  - Tokai University Hospital, Isehara
  - Shimane University Hospital, Izumo
  - Kurume University Hospital, Kurume
  - Nagoya University Hospital, Nagoya
  - Okayama University Hospital, Okayama
  - Kansai Electric Power Hospital, Osaka
  - Shiga University of Medical Science Hospital, Ōtsu
  - Toranomon Hospital, Tokyo
  - Juntendo University Hospital, Tokyo
  - The University of Tokyo Hospital, Tokyo
  - National Center for Global Health and Medicine, Tokyo
  - Tokyo-Eki Center-building Clinic, Tokyo, Chuo-ku
- Malaysia (24):
  - Hospital Ampang, Ampang
  - Hospital Selayang, Batu Caves
  - Hospital Sultanah Nora Ismail, Batu Pahat
  - Hospital Pulau Pinang-Pulau Pinang-21953, George Town
  - Hospital Raja Permaisuri Bainun, Ipoh
  - Hospital Sultanah Aminah, Johor Bahru
  - Hospital Kajang, Kajang, Selangor
  - Hospital Tengku Ampuan Rahimah, Klang
  - Hospital Raja Perempuan Zainab II, Kota Bharu
  - Hospital Queen Elizabeth, Kota Kinabalu
  - Hospital Kuala Lumpur, Kuala Lumpur
  - University of Malaya Medical Centre, Kuala Lumpur
  - Hospital Tuanku Ampuan Najihah, Kuala Pilah
  - Hospital Tengku Ampuan Afzan, Kuantan
  - Hospital Umum Sarawak, Kuching
  - Hospital Kulim, Kulim
  - Hospital Melaka, Malacca
  - Hospital Pakar Sultanah Fatimah, Muar town
  - Hospital Seberang Jaya, Perai
  - Hospital Sultan Abdul Aziz Shah, Serdang
  - Hospital Tuanku Ja'afar, Seremban
  - Hospital Taiping, Taiping
  - Hospital Teluk Intan, Teluk Intan
  - Hospital Sultan Haji Ahmad Shah, Temerluh
- Mexico (5):
  - Instituto de investigación aplicado a la neurociencia, Durango
  - Centro de Investigacion Clinica y Medicina Traslacional (CIMeT), Guadalajara
  - Instituto Nacional de Cardiologia Ignacio Chavez, Mexico City
  - Merida Investigación Clínica, Mérida
  - FAICIC S de RL de C.V., Veracruz
- New Zealand (3):
  - Auckland City Hospital, Auckland
  - North Shore Hospital, Auckland, Takapuna
  - Taranaki Base Hospital, New Plymouth
- Portugal (10):
  - ULS da Região de Aveiro, Aveiro
  - CHUC - Centro Hospitalar e Universitário de Coimbra, EPE, Coimbra
  - Unidade Local de Saúde do Algarve, E.P.E, Faro
  - SESARAM, Funchal
  - ULS de São José, Lisbon
  - Unidade Local de Saúde Santa Maria, Lisbon
  - Hospital Beatriz Ângelo, Loures
  - Centro Hospitalar Universitário São João,EPE, Porto
  - Unidade Local de Saúde de Matosinhos, Senhora da Hora
  - Unidade Local De Saude Da Arrabida E.P.E., Setúbal
- South Korea (18):
  - Korea University Ansan Hospital, Ansan-si
  - Pusan National University Hospital, Busan
  - Soon Chun Hyang University Hospital Cheonan, Cheonan-si
  - Chungbuk National University Hospital, Cheongju-si
  - Kyungpook National University Hospital, Daegu
  - Keimyung University Dongsan Hospital, Deagu
  - Inje University Ilsan Paik Hospital, Goyang-si
  - Hanyang University Guri Hospital, Guri-si
  - Chung-Ang University Gwangmyeong Hospital, Gwangmyeong
  - The Catholic University of Korea, Incheon St. Mary's Hospital, Incheon
  - CHA Bundang Medical Center, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - The Catholic University of Korea, Yeouido St.Mary's Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju
- Taiwan (16):
  - E-Da Hospital, Kaohsiung City
  - Lotung Poh-Ai Hospital, Luodong Township
  - Taipei Medical University-Shuang Ho Hospital, New Taipei City
  - Fu Jen Catholic University Hospital, New Taipei City
  - Chung Shan Medical University Hospital, Taichung
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Tungs' Taichung MetroHarbor Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Hospital, Liouying, Tainan
  - MacKay Memorial Hospital, Taipei
  - Cathay General Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Shin Kong Wu Ho-Su Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Taipei Municipal Wanfang Hospital, Taipei
- United Kingdom (39):
  - Antrim Area Hospital, Antrim
  - Basildon Hospital, Basildon
  - South Eastern Health & Social Care Trust, Belfast
  - Belfast Health and Social Care Trust, Belfast
  - Oakenhurst Medical Practice, Blackburn
  - University Hospitals Sussex NHS Foundation Trusts, Brighton
  - Southmead Hospital, Bristol
  - Coniston Medical Practice, Bristol
  - West Suffolk NHS Foundation Trust, Bury St Edmunds
  - Broomfield Hospital, Chelmsford
  - Hathaway Medical Centre, Chippenham
  - Clevedon Medical Centre, Clevedon
  - Queen Alexandra Hospital, Cosham
  - Daisy Hill Hospital, County Down
  - University Hospitals Coventry and Warwickshire NHS Trust, Coventry
  - Orchard Court Surgery, Darlington
  - Dorset County Hospital NHS Foundation Trust, Dorset
  - Highland Clinical Research Facility, Fulwood
  - Gloucestershire Royal Hospital, Gloucester
  - James Paget University Hospital, Great Yarmouth
  - Hereford County Hospital, Hereford
  - Ipswich Hospital (UK), Ipswich
  - St Luke's Hospital, Little Horton Lane
  - Aintree University Hospital, Liverpool
  - King's College Hospital, London
  - St George's University Hospitals NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - Altnagelvin Area Hospital, Londonderry
  - Norfolk and Norwich University Hospital, Norfolk
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Banbury Cross Health Centre, Oxford
  - Churchill Hospital, Oxford
  - Pickering Medical Practice, Pickering
  - Royal Berkshire Hospital, Reading
  - Alexandra Hospital, Redditch
  - The Royal Shrewsbury Hospital, Shrewsbury
  - Lister Hospital, Stevenage
  - Great Western Hospital, Swindon
  - Royal Cornwall Hospital, Truro

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.clinicalstudies.boehringer-ingelheim.com/msw/datatransparency